CLINICAL TRIAL: NCT02452463
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled Study Evaluating Nintedanib Versus Placebo as Prophylaxis Against Radiation Pneumonitis in Patients With Unresectable NSCLC Undergoing Chemoradiation Therapy
Brief Title: Nintedanib Compared With Placebo in Treating Against Radiation-Induced Pneumonitis in Patients With Non-small Cell Lung Cancer That Cannot Be Removed by Surgery and Are Undergoing Chemoradiation Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: I 257814; NCI-2015-00704 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 257814 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-03

CONDITIONS: Lung Non-Squamous Non-Small Cell Carcinoma; Radiation-Induced Pneumonitis; Stage II Lung Non-Small Cell Cancer AJCC v7; Stage IIA Lung Non-Small Cell Carcinoma AJCC v7; Stage IIB Lung Non-Small Cell Carcinoma AJCC v7; Stage III Lung Non-Small Cell Cancer AJCC v7; Stage IIIA Lung Non-Small Cell Cancer AJCC v7; Stage IIIB Lung Non-Small Cell Cancer AJCC v7; Stage IV Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Radiation Pneumonitis; Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Immunoglobulin G; Disulfides; nintedanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (nintedanib) (Experimental): Beginning 4-8 weeks after completion of radiation therapy, patients receive nintedanib PO BID on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nintedanib; Procedure: Quality-of-Life Assessment
- Arm II (placebo) (Placebo Comparator): Beginning 4-8 weeks after completion of radiation therapy, patients receive placebo capsules PO BID on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Placebo; Procedure: Quality-of-Life Assessment
- Arm III (nintedanib, durvalumab) (Experimental): Beginning 4-8 weeks after completion of radiation therapy, patients receive nintedanib PO BID on days 1-28 and standard of care durvalumab IV over 60 minutes on days 1 and 15. Treatment with nintedanib repeats every 28 days for up to 6 cycles and treatment with durvalumab repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Drug: Nintedanib; Procedure: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
  Arms: Arm III (nintedanib, durvalumab)
Drug: Nintedanib — Given PO
  Other Names: BIBF 1120; BIBF-1120; Intedanib; Multitargeted Tyrosine Kinase Inhibitor BIBF 1120; tyrosine kinase inhibitor BIBF 1120; Vargatef
  Arms: Arm I (nintedanib); Arm III (nintedanib, durvalumab)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This trial studies the side effects and how well nintedanib works compared to a placebo in treating against radiation-induced pneumonitis (inflammation of the lungs) in patients with non-small cell lung cancer that cannot be removed by surgery and are undergoing chemoradiation therapy. Nintedanib may help shrink or slow the growth of radiation-induced pneumonitis by blocking some of the enzymes needed for cells to grow and may prevent the growth of new blood vessels. It may also help reduce the recurrence of non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of the combination of durvalumab with nintedanib in patients with unresectable Stage II/III/oligometastatic IV non-small cell lung carcinoma (NSCLC). (Phase I) II. To compare the rate of symptomatic radiation pneumonitis at 6 months after completion of chemoradiation in patients with unresectable stage II/III/ oligometastatic IV NSCLC who completed chemoradiation followed by nintedanib versus placebo. (Phase II)

SECONDARY OBJECTIVES:

I. To compare the quality of life (QOL) in patients who received nintedanib versus placebo during active treatment until 6 months after completion of treatment.

II. To compare the progression-free survival, overall survival and 1-year progression-free survival rate in patients who received nintedanib versus placebo.

III. To compare pulmonary function test (PFT) results and radiation pneumonitis (RP) score in patients who received nintedanib versus placebo.

IV. To compare the composite index (based on PFT, RP score and QOL) at the end of active treatment and 6 months after completion of treatment between patients who received nintedanib versus placebo.

EXPLORATORY OBJECTIVES:

I. To investigate blood-based biomarkers in evaluating risk of developing radiation pneumonitis as well as the efficacy of nintedanib.

OUTLINE: This is a phase I, dose-escalation study of nintedanib followed by a phase II study. Patients who are not receiving durvalumab as standard of care prior to establishment of the recommended phase II dose are randomized to 1 of 2 arms. Patients receiving durvalumab are assigned to Arm III.

ARM I: Beginning 4-8 weeks after completion of radiation therapy, patients receive nintedanib orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Beginning 4-8 weeks after completion of radiation therapy, patients receive placebo capsules PO BID on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

ARM III: Beginning 4-8 weeks after completion of radiation therapy, patients receive nintedanib PO BID on days 1-28 and standard of care durvalumab intravenously (IV) over 60 minutes on days 1 and 15. Treatment with nintedanib repeats every 28 days for up to 6 cycles and treatment with durvalumab repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, between 76-97 days, between 166-187 days, and then between 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-proven non squamous cell NSCLC; mixed histology with small cell lung carcinoma (SCLC) component not allowed
* Patients with stage II ? IV non squamous cell NSCLC who received at least 54 Gy of total planned thoracic radiation dose will be eligible; patients must have received at least one cycle of chemotherapy concurrently during the course of thoracic radiation; regimens allowed are platinum combinations with either etoposide or a taxane regardless of histology subtype; platinum with pemetrexed for patients with non-squamous NSCLC only; patients with oligometastatic stage IV cancer are eligible if they have received only one line of systemic therapy for their stage IV cancer prior to the concurrent chemoradiation phase
* Patient must have had a complete response (CR)/partial response (PR)/stable disease (SD), 4-6 weeks after completing last fraction of radiation therapy
* Eastern Cooperative Oncology Group (ECOG) performance score 0-2
* Absolute neutrophil count (ANC) >= 1,500/uL
* Platelet count >= 100,000/uL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< normal or for those with Gilbert?s syndrome =< 1.5 times upper limit of normal (ULN) OR direct bilirubin normal (per institute standards)
* Aspartate aminotransferase (AST) =< 1.5 x ULN; alanine aminotransferase (ALT) and AST =< 2.5 x ULN is acceptable if there is liver metastasis
* Fertile patients must use adequate contraception

Exclusion Criteria:

* Whole-brain radiotherapy (WBRT) < 14 days from the anticipated start of nintedanib/placebo administration
* Squamous cell NSCLC
* Unable to start nintedanib/placebo treatment between 4-8 weeks after completing the last dose of thoracic radiation
* Active untreated brain or leptomeningeal metastases; in patients with treated central nervous system (CNS) metastases, eligible if symptoms controlled for at least 4 weeks; dexamethasone allowed if total daily dose does not exceed 2 mg
* Major injuries or surgery (e.g., craniotomy) < 28 days from the start of nintedanib/placebo administration; wound should be healed prior to starting therapy
* Second malignancies are allowed as long as the disease does not require active treatment with concomitant systemic cytotoxic chemotherapy, investigational or biologic therapy (e.g., anti-cytotoxic T-lymphocyte-associated protein 4 [CTLA4] or human epidermal growth factor receptor 2 [HER2] monoclonal antibodies); hormone-related therapies (e.g., gonadotrophin releasing hormone (LHRH) agonists, tamoxifen, etc.) are allowed
* Concurrent uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would increase the risk associated with study participation and/or limit compliance with study requirements
* Inability to swallow study medication
* Presence of active malabsorption disorder (e.g., flare episodes documented within the preceding 3 months, presence of symptoms requiring daily medications for control) or history of extensive small bowel resection
* Known bleeding or thrombotic diathesis
* History of arterial or venous thromboembolic event within 12 months prior to study participation
* Active hemoptysis or history of clinically relevant hemoptysis as determined by the treating physician; patients who had history of transient minor hemoptysis after bronchoscopic biopsy are eligible unless deemed otherwise by the treating physician
* Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or higher proteinuria
* Investigational agent administered < 28 days prior to treatment with nintedanib. Last dose of systemic chemotherapy administered < 14 days prior to treatment with nintedanib
* Known chronic active hepatitis B or hepatitis C; human immunodeficiency virus (HIV)-positive patients receiving or are candidates for antiretroviral therapy are also excluded
* Pregnancy or breast feeding; female patients with child-bearing potential must have a negative pregnancy test (beta-human chorionic gonadotropin [B-HCG] test in urine or serum) prior to commencing study treatment
* Creatinine > 1.5 x ULN or creatinine clearance levels (CrCL) < 45 mL/min
* Centrally located tumors with radiographic evidence (computed tomography [CT] or magnetic resonance imaging [MRI]) of local invasion of major blood vessels
* Therapeutic anticoagulation (except low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous devise) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid < 325 mg per day)
* Active or previous autoimmune disease requiring treatment within the past 2 years will exclude patients from receiving immune checkpoint inhibitor in this study. Exception allowed: endocrine conditions treated with necessary hormone replacement or other supportive medication; vitiligo, alopecia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace K Dy, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Rimner A, Moore ZR, Lobaugh S, Geyer A, Gelblum DY, Abdulnour RE, Shepherd AF, Shaverdian N, Wu AJ, Cuaron J, Chaft JE, Zauderer MG, Eng J, Riely GJ, Rudin CM, Els NV, Chawla M, McCune M, Li H, Jones DR, Sopka DM, Simone CB 2nd, Mak R, Weinhouse GL, Liao Z, Gomez DR, Zhang Z, Paik PK. Randomized Phase 2 Placebo-Controlled Trial of Nintedanib for the Treatment of Radiation Pneumonitis. Int J Radiat Oncol Biol Phys. 2023 Aug 1;116(5):1091-1099. doi: 10.1016/j.ijrobp.2023.02.030. Epub 2023 Mar 7. PMID 36889516

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in the "Arm III (Nintedanib, Durvalumab)" Arm - study closed prior to any patients being enrolled in this arm.
Period: Overall Study
Arm/Group | Arm I (Nintedanib) | Arm II (Placebo) | Arm III (Nintedanib, Durvalumab)
Started | 5 | 3 | 0 (No participants were enrolled in the "Arm III (Nintedanib, Durvalumab)" Arm.)
Completed | 3 | 1 | 0
Not Completed | 2 | 2 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Study Suspended | 1 | 0 | 0
Not completed — Recommended by DSMB | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated prior to enrollment in Arm 3.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Nintedanib) | Arm II (Placebo) | Arm III (Nintedanib, Durvalumab) | Total
Number analyzed (Participants) | 5 | 3 | 0 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.40 (5.94) | 68.00 (4.58) |  | 65.75 (5.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 |  | 5
  Male | 1 | 2 |  | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 0 |  | 0
  White | 5 | 3 |  | 8
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 |  | 8
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 21.75 (5.47) | 32.15 (3.84) |  | 25.65 (7.09)
Chemotherapy [Count of Participants; unit: Participants]
  CARBOPLATIN + PACLITAXEL (TAXOL) | 2 | 1 |  | 3
  CARBOPLATIN + PEMETREXED | 1 | 2 |  | 3
  CISPLATIN + ETOPOSIDE (VP-16) | 1 | 0 |  | 1
  CISPLATIN + PEMETREXED | 1 | 0 |  | 1
Smoking Status [Count of Participants; unit: Participants]
  Current | 2 | 1 |  | 3
  Former | 2 | 2 |  | 4
  Unknown | 1 | 0 |  | 1
Force Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: Percentage of Predicted FEV1] | 66.70 (29.59) | 72.67 (6.81) |  | 68.94 (22.87)
Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: Percentage of Predicted FVC] | 91.72 (26.74) | 82.93 (5.97) |  | 88.43 (20.96)
Diffusing Capacity for Carbon Monoxide (DLCO) [Mean (Standard Deviation); unit: Percentage of Predicted DLCO] | 60.52 (27.21) | 77.93 (10.04) |  | 67.05 (23.09)
peak expiratory flow (PEF) [Mean (Standard Deviation); unit: Percentage of Predicted PEF] | 67.22 (33.78) | 74.90 (15.89) |  | 70.10 (27.20)
total lung capacity (TLC) [Mean (Standard Deviation); unit: Percentage of Predicted TLC] | 110.60 (18.29) | 99.17 (8.96) |  | 106.31 (15.78)
Eastern Cooperative Oncology Group Performance Status(ECOG) [Count of Participants; unit: Participants] — 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    Fully active | 3 | 0 |  | 3
    Restricted in physically strenuous activity | 2 | 3 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Portion of Common Terminology Criteria for Adverse Events Grade 2 or Higher Radiation Pneumonitis
Description: Will compare the rate of symptomatic radiation pneumonitis in patients who received nintedanib versus placebo. Assessed using the intent-to-treat principle and a one-sided exact test about the Cochran-Mantel-Haenszel correlation and regression test.
  The grade 2 or higher radiation penumonitis is identified by the Common Terminology Criteria for Adverse Events.
Time Frame: At 6 months after completion of chemoradiation
Population: Study was terminated prior to enrollment in Arm 3.
Measure: Number; unit: proportion of participants
Arm/Group | Arm I (Nintedanib) | Arm II (Placebo) | Arm III (Nintedanib, Durvalumab)
Number analyzed (Participants) | 5 | 3 | 0
proportion of participants | 0.00 | 0.67 |
Statistical Analysis 1: Comparison: Arm I (Nintedanib) vs Arm II (Placebo); Test type: Superiority; p = 0.107, Cochran-Mantel-Haenszel

2. Secondary Outcome: Number of Participants With Adverse Events, Graded According to Common Terminology Criteria for Adverse Events Version 4.0
Description: The frequency of toxicities will be tabulated by grade.
Time Frame: Up to 2.5 years post-treatment
Population: Study was discontinued prior to subjects being enrolled in Arm III
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nintedanib) | Arm II (Placebo) | Arm III (Nintedanib, Durvalumab)
Number analyzed (Participants) | 5 | 3 | 0
Participants
  Grade 1 Maximum AE | 2 | 0 | 0
  Grade 2 Maximum AE | 1 | 1 | 0
  Grade 3 Maximum AE | 1 | 0 | 0
  No Treatmetn Related AE | 1 | 2 | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival will be reported using standard Kaplan-Meier methods. Comparisons of overall survival between study arms may utilize the two-sided stratified log-rank test.
Time Frame: 1 year survival, with follow-up assessed up to 2.5 years post-treatment
Population: Study was terminated prior to enrollment in Arm 3.
Measure: Number (95% Confidence Interval); unit: Percent survival at 1 year
Arm/Group | Arm I (Nintedanib) | Arm II (Placebo) | Arm III (Nintedanib, Durvalumab)
Number analyzed (Participants) | 5 | 3 | 0
Percent survival at 1 year | 53.0 [7.0 to 86.0] | 100.0 [100.0 to 100.0] |
Statistical Analysis 1: Comparison: Arm I (Nintedanib) vs Arm II (Placebo); Null Hypotheses: OS distributions are equal; Test type: Superiority; p = 0.75, Log Rank

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival will be reported using standard Kaplan-Meier methods. Comparisons of progression-free survival between study arms may utilize the two-sided stratified log-rank test.
Time Frame: 1 year progression-free survival, with follow-up assessed up to 2.5 years post-treatment
Population: Study was terminated prior to enrollment in Arm 3.
Measure: Number (95% Confidence Interval); unit: Percent survival at 1 year
Arm/Group | Arm I (Nintedanib) | Arm II (Placebo) | Arm III (Nintedanib, Durvalumab)
Number analyzed (Participants) | 5 | 3 | 0
Percent survival at 1 year | 25.0 [1.0 to 67.0] | 100.0 [100.0 to 100.0] |
Statistical Analysis 1: Comparison: Arm I (Nintedanib) vs Arm II (Placebo); Null Hypotheses: PFS distributions are equal; Test type: Superiority; p = 0.25, Log Rank

5. Secondary Outcome: Percent Changes in Overall Quality of Life and Symptom Scores
Description: Percent changes in the quality of life and symptom scores may be compared between study arms using the Wilcoxon rank sum or independent sample t-tests, as appropriate.
  The quality of life scores are obtained using the Lung Cancer Symptom Scale (LCSS) The scores range from 0 to 68, where 0 indicates poor quality of life and 68 indicates good quality of life. The percent change from baseline was calculated as 100*(post treatment - baseline) / baseline.
Time Frame: Baseline up to 2.5 years post-treatment
Population: Study was terminated prior to enrollment in Arm 3. For Arms 1 and 2, not all follow-up tests were completed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm I (Nintedanib) | Arm II (Placebo) | Arm III (Nintedanib, Durvalumab)
Number analyzed (Participants) | 2 | 2 | 0
percent change | 110.00 (70.71) | -16.35 (12.24) |
Statistical Analysis 1: Comparison: Arm I (Nintedanib) vs Arm II (Placebo); Test type: Superiority; p = 0.131, t-test, 2 sided

6. Secondary Outcome: Percent Change in Pulmonary Function Tests
Description: Percent change in pulmonary function test, relative to baseline, will be evaluated within each study arm using the Wilcoxon signed rank or paired t-tests, as appropriate. Changes in pulmonary function tests may be compared between study arms using the Wilcoxon rank sum or independent sample t-tests, as appropriate.
Time Frame: Baseline up to 2.5 years post-treatment
Population: Study was terminated prior to enrollment in Arm 3. For Arms 1 and 2, not all follow-up tests were completed.
Measure: Mean (Standard Deviation); unit: percent of change
Arm/Group | Arm I (Nintedanib) | Arm II (Placebo) | Arm III (Nintedanib, Durvalumab)
Number analyzed (Participants) | 2 | 2 | 0
percent of change | -28.29 (13.43) | 11.02 (8.59) |
Statistical Analysis 1: Comparison: Arm I (Nintedanib) vs Arm II (Placebo); Test type: Superiority; p = 0.073, t-test, 2 sided

7. Secondary Outcome: Changes in Radiation Pneumonitis Scores
Description: Changes in radiation pneumonitis scores, relative to baseline, will be evaluated within each study arm using the Wilcoxon signed rank or paired t-tests, as appropriate. Changes in radiation pneumonitis scores may be compared between study arms using the Wilcoxon rank sum or independent sample t-tests, as appropriate.
  The radiation pneumonitis scores were obtained using semi quantitative analysis will be performed for the presence of ground-glass opacity, consolidation, reticulation, mosaic perfusion, traction bronchiectasis and honeycombing for each lung zone and scored on a four point scale (0 = no involvement, 1 ≤ 25%; 2 = 26 50%; 3 = 51 75% and 4 ≥ 76%). The scores are averaged across two radiologists.
Time Frame: Baseline up to 2.5 years post-treatment
Population: Study was terminated prior to enrollment in Arm 3. For Arms 1 and 2, not all follow-up tests were completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Nintedanib) | Arm II (Placebo) | Arm III (Nintedanib, Durvalumab)
Number analyzed (Participants) | 4 | 2 | 0
score on a scale | 0.50 (0.58) | 0.75 (0.35) |
Statistical Analysis 1: Comparison: Arm I (Nintedanib) vs Arm II (Placebo); Test type: Superiority; p = 0.616, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm I (Nintedanib); Comparing change relative to baseline; Test type: Superiority; p = 0.183, Paired T-test
Statistical Analysis 3: Comparison: Arm II (Placebo); Evaluating change relative to baseline; Test type: Superiority; p = 0.203, paired T-test

8. Secondary Outcome: Responses Rates
Description: Complete response and complete/partial response rates will be reported by study arm and chemotherapy regimen using Wilson 95% confidence intervals. The responses rates will be compared between study arms using the Cochran-Mantel-Haenszel exact test.
  The objective tumor response was assessed using RECIST 1.1:
  1. Complete Response (CR): Disappearance of all target lesions. Any lymph nodes must have a reduction in short axis to < 10 mm.
  2. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  3. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions. The appearance of one or more new lesions is also considered progression.
  4. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameter while on study.
  Overall response = CR + PR.
Time Frame: Up to 2.5 years post-treatment
Population: Study was terminated prior to enrollment in Arm 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nintedanib) | Arm II (Placebo) | Arm III (Nintedanib, Durvalumab)
Number analyzed (Participants) | 5 | 3 | 0
Participants
  SD/PD | 5 | 3 |
  CR/PR | 0 | 0 |
Statistical Analysis 1: Comparison: Arm I (Nintedanib) vs Arm II (Placebo); Test type: Superiority; p = 1.00, Cochran-Mantel-Haenszel

9. Secondary Outcome: Biomarker Analysis
Description: The tethered cationic lipoplex nanoparticle biochip, microfluidic cationic lipoplex nanoparticle biochip and real-time quantitative reverse transcription-polymerase chain reaction measurements for the expression of micro ribonucleic acid -1, -21, -127 and -155 will be made. The micro ribonucleic acid expressions, vitamin D levels, and mitochondrial deoxyribonucleic acid levels will be treated as continuous and reported by radiation pneumonitis status using the mean, median and standard deviation. Comparisons will be made between groups using a two-sided permutation t-test.
Time Frame: Up to 97 days post-treatment
Population: Due to early termination of the study, the biomarker data was never collected and analyzed.
Arm/Group | Arm I (Nintedanib) | Arm II (Placebo) | Arm III (Nintedanib, Durvalumab)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start date of intervention until 30 days after the last treatment intervention, up to 2.5 years.
Description: All treated patients in Arms I and II.
  No participants were enrolled in the "Arm III (Nintedanib, Durvalumab)" Arm, therefore no adverse events are reported.
Arm/Group | Arm I (Nintedanib) | Arm II (Placebo) | Arm III (Nintedanib, Durvalumab)
All-Cause Mortality (participants affected / at risk) | 2/5 | 1/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Nintedanib) (N=5) | Arm II (Placebo) (N=3) | Arm III (Nintedanib, Durvalumab) (N=0)
Lung infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Nintedanib) (N=5) | Arm II (Placebo) (N=3) | Arm III (Nintedanib, Durvalumab) (N=0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (4) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT02452463/Prot_SAP_000.pdf